CLINICAL TRIAL: NCT00878553
Title: A Phase 2, Double-Blind, Placebo-Controlled, Double-Dummy, Cross-Over Study to Investigate the Hypnotic Activity of Three Doses (10mg, 15mg, 20mg) of a New Zaleplon Prototype, SKP-1041, in Adults With Primary Insomnia
Brief Title: Study of Sleep-maintenance Activity of 3 Doses of SKP-1041
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Somnus Therapeutics, Inc. (Industry)
Collaborators: INC Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SOM201
Record Dates: First submitted 2009-03-19; First posted 2009-04-09 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Sleep Disorder; Primary Insomnia
Keywords: insomnia; middle of the night; sleep maintenance
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Sugars; zaleplon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Two placebo tablets administered orally at bedtime for two consecutive nights to each patient per crossover randomized sequence
  Interventions: Drug: placebo
- 10 mg SKP-1041 (Experimental): One 10 mg SKP-1041 controlled release zaleplon tablet plus one placebo tablet administered orally at bedtime for two consecutive nights to each patient per crossover randomized sequence
  Interventions: Drug: SKP-1041 (experimental formulation of zaleplon)
- 15 mg SKP-1041 (Experimental): One 15 mg SKP-1041 controlled release zaleplon tablet plus one placebo tablet administered orally at bedtime for two consecutive nights to each patient per crossover randomized sequence
  Interventions: Drug: SKP-1041 (experimental formulation of zaleplon)
- 20 mg SKP-1041 (Experimental): Two 10 mg SKP-1041 controlled release zaleplon tablets administered orally at bedtime for two consecutive nights to each patient per crossover randomized sequence
  Interventions: Drug: SKP-1041 (experimental formulation of zaleplon)

INTERVENTIONS:
Drug: placebo — tablet at bedtime
  Other Names: sugar pill
  Arms: Placebo
Drug: SKP-1041 (experimental formulation of zaleplon) — tablet at bedtime
  Other Names: zaleplon
  Arms: 10 mg SKP-1041; 15 mg SKP-1041; 20 mg SKP-1041

SUMMARY:
SKP-1041 is a new formulation of a marketed sleeping agent called zaleplon. Zaleplon is currently available as Sonata as well as several generic formulations. Sonata and its generics induce sleep soon after ingestion. SKP-1041, however, is a formulation that is designed to become active 2-3 hours after ingestion. It is intended for use in people who have no trouble falling to sleep but who often awaken in the middle of the night. This trial will determine the best dose to prevent those awakenings.

DETAILED DESCRIPTION:
Patients will participate in the study for approximately 44 to 56 days, including a 14- to 21-day Screening Period, 4 Treatment Periods each followed by washout periods, and a final Follow-up Visit. Patients will receive their randomly assigned study medication and spend 2 nights in a sleep laboratory, subsequently returning home for a 4- to 7-day washout period between each treatment period. The fourth and final treatment period will include a third night at the site during which all patients will continue to receive the same study medication as on the first 2 nights of this treatment period. Blood will be drawn from all patients for pharmacokinetic analyses at specific time intervals. Patients will undergo final safety assessments 2 to 5 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Primary insomnia characterized by chronic difficulty maintaining sleep

Exclusion Criteria:

* History of restless legs syndrome, sleep apnea, narcolepsy, or parasomnias;
* Any clinically relevant acute or chronic diseases which could interfere with the patient's safety during this trial or with this tablet's absorption;
* Pregnancy;
* History of medication allergies;
* Use of medication that might interfere with this study;
* Recent travel across more than 3 time zones.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Freeman, PhD, Principal Investigator — Clinilabs, Inc.; Steven G. Hull, MD, Principal Investigator — Vince and Associates Clinical Research; Russell Rosenberg, PhD, Principal Investigator — Neurotrials Inc.; James K. Walsh, PhD, Principal Investigator — Sleep Medicine and Research Center; David J. Seiden, MD, Principal Investigator — Broward Research Group; Helene A. Emsellem, MD, Principal Investigator — Emsellem MD PC; D. Alan Lankford, PhD, Principal Investigator — Sleep Disorders Center of Georgia; Beth E. Safirstein, MD, Principal Investigator — MD Clinical

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 394 potential patients were screened by 8 U.S. investigative sites for enrollment into this study. Of these potential patients, 327 failed to complete the screening process.
Pre-assignment Details: 5 of the 67 patients who were enrolled and randomized into this crossover sleep study did not complete it. The reasons for discontinuation were withdrawal of consent (2 patients), automobile accident(1), family emergency (1) and lost to follow up(1). One additional patient withdrew after completing the sleep study but prior to the PK substudy.
Groups:
- Baseline: All Randomized Patients: The second screening visit consisted of 2 consecutive sleep laboratory nights of placebo pretreatment and full PSG recordings. The 67 patients who met entry criteria were then randomized to four treatment sequences with their screening night mean PSG parameters defined as their baseline.
  This trial was comprised of 2 study periods: Sleep and Pharmacokinetic (PK). Each of 67 patients was randomly assigned a sequence of the four treatment arms, washed out, and then crossed over to the next assigned treatment in their sequence for the Sleep Study. For each of these treatment arms, two "double-dummy" tablets were administered at bedtime for two consecutive nights. An additional (third) dosing night allowed for pharmacokinetic characterization of the investigational zaleplon formulation. In this PK Substudy, patient's plasma concentrations were measured after a single dose in parallel group design.
- Placebo (Sugar Pill): Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive placebo treatment. Two placebo tablets were administered orally at bedtime for two consecutive nights during the Sleep Study, after which patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned for the next treatment in their randomized sequence.
- 10 mg SKP-1041: Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive 10mg of the investigational zaleplon delayed and sustained release SKP-1041 tablets. One 10 mg SKP-1041 tablet and one placebo tablet were administered orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
- 15 mg SKP-1041: Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive 15mg of the investigational zaleplon delayed and sustained release SKP-1041 tablets. One 15 mg SKP-1041 tablet and one placebo tablet were administered orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
- 20 mg SKP-1041: Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive 20mg of the investigational zaleplon delayed and sustained release SKP-1041 tablets. Two 10 mg SKP-1041 tablets were administered orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
Period: Sleep Study
Arm/Group | Baseline: All Randomized Patients | Placebo (Sugar Pill) | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Started | 67 (This Intention to Treat population includes all randomized patients; one dropped prior to treatment.) | 0 | 0 | 0 | 0
Number of Patients Receiving Placebo | 66 | 0 | 0 | 0 | 0
Number of Patients Receiving 10mg | 65 | 0 | 0 | 0 | 0
Number of Patients Receiving 15mg | 65 | 0 | 0 | 0 | 0
Number of Patients Receiving 20mg | 65 | 0 | 0 | 0 | 0
Completed | 62 (5 patient withdraws result in greater than 5 lost patient data across groups due to CROSSOVER design) | 0 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — car accident | 1 | 0 | 0 | 0 | 0
Not completed — family emergency | 1 | 0 | 0 | 0 | 0
Period: PK Study
Arm/Group | Baseline: All Randomized Patients | Placebo (Sugar Pill) | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Started | 0 (A total of 62 randomized patients started this parallel group, single dose PK substudy.) | 16 (During the PK period, 16 randomized participants received one bedtime dose of SKP-1041 placebo.) | 17 (During the PK period, 17 randomized participants received one bedtime dose of 10mg SKP-1041.) | 14 (During the PK period, 14 participants were randomized to receive one bedtime dose of 15mg SKP-1041.) | 15 (During the PK period, 15 randomized participants received one bedtime dose of 20mg SKP-1041.)
Completed | 0 (A total of 61 randomized patients completed this parallel group, single dose PK substudy.) | 16 | 17 | 13 (One patient withdrew consent after completing the Sleep Substudy and prior to starting PK substudy.) | 15
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: 10mg SKP-1041, 15mg SKP-1041, Placebo, 20mg SKP-1041
- Sequence 2: Placebo, 10mg SKP-1041, 20mg SKP-1041, 15mg SKP-1041
- Sequence 3: 20mg SKP-1041, Placebo, 15mg SKP-1041, 10mg SKP-1041
- Sequence 4: 15mg SKP-1041, 10mg SKP-1041, 20mg SKP-1041, Placebo
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 16 | 17 | 17 | 17 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 17 | 17 | 67
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.3 (9.94) | 47.1 (9.23) | 42.5 (11.95) | 47.5 (9.47) | 46.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 8 | 8 | 41
  Male | 5 | 3 | 9 | 9 | 26
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 17 | 17 | 67

OUTCOME MEASURES:

1. Primary Outcome: Wake After Sleep Onset During Hours 3 to 7 Post-dose (WASO 3-7)
Description: Wake time After Sleep Onset hours 3-7 Pairwise comparisons of treatment group vs. placebo mean change from baseline in minutes per polysomnographic recording. Each patient receives baseline placebo and then each treatment dose at bedtime for two nights of sleep laboratory PSG measurements. The WASO3-7 mean of each two night visit is then used to compare placebo vs. treatment change from baseline minutes awake during hours 3 through 7 post-dose.
Time Frame: Hours 3-7 (inclusive) after tablet ingestion
Population: Efficacy analyses were performed on the Intention to Treat Population(all randomized patients).
Measure: Mean (Standard Error); unit: minutes
Groups:
- Placebo (Sugar Pill): Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive placebo treatment in place of the investigational zaleplon delayed and sustained release SKP-1041 tablets. These patients received two placebo tablets orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
Arm/Group | Placebo (Sugar Pill) | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 67 | 67 | 67 | 67
minutes | -40.19 (2.385) | -48.79 (2.420) | -50.17 (2.421) | -49.34 (2.422)
Statistical Analysis 1: Comparison: Placebo (Sugar Pill) vs 10 mg SKP-1041; Literature-based estimates of WASO (Wake After Sleep Onset) SD (Standard Deviation) range from 39 to 45 minutes. Null hypothesis: difference between mean WASO3-7 values for placebo and the 15-mg SKP-1041 dose level equals 0. By using a 2-sided, 1-sample t test at the 5% level of significance of this null hypothesis and an assumed SD of 45 minutes, a sample size of 54 completed patients was calculated to provide 90% power to detect a mean treatment difference of 20 minutes; Test type: Superiority or Other; p = 0.0118, Mixed Models Analysis — Change from baseline in mean WASO3-7 compared values for the 20-mg dose vs. placebo. If that comparison demonstrated superiority of the 20-mg dose, then results for the 15-mg dose vs. placebo were compared; if significant, then 10-mg vs. placebo; This hierarchical, 2-sided testing procedure maintained the overall level of significance at approximately 0.05; Mean Difference (Net) = -8.606, 95% CI 2-sided [-15.284 to -1.927], Standard Error of Mean 2.420 — Adjusted mean differences were analyzed via general linear model that used change from baseline as response variable and included effects for patient, period, sequence, and treatment. A negative mean change from baseline indicates an improvement
Statistical Analysis 2: Comparison: Placebo (Sugar Pill) vs 15 mg SKP-1041; Literature-based estimates of WASO SD range from 39 to 45 minutes. Null hypothesis: difference between mean WASO3-7 values for placebo and the 15-mg SKP-1041 dose level equals 0. By using a 2-sided, 1-sample t test at the 5% level of significance of this null hypothesis and an assumed SD of 45 minutes, a sample size of 54 completed patients was calculated to provide 90% power to detect a mean treatment difference of 20 minutes; Test type: Superiority or Other; p = 0.0037, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; This hierarchical, 2-sided testing procedure maintained the overall level of significance at approximately 0.05; Mean Difference (Net) = -9.98, 95% CI 2-sided [-16.685 to -3.275], Standard Error of Mean 2.421 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo (Sugar Pill) vs 20 mg SKP-1041; Literature-based estimates of WASO SD range from 39 to 45 minutes. Null hypothesis: difference between mean WASO3-7 values for placebo and the 20-mg SKP-1041 dose level equals 0. By using a 2-sided, 1-sample t test at the 5% level of significance of this null hypothesis and an assumed SD of 45 minutes, a sample size of 54 completed patients was calculated to provide 90% power to detect a mean treatment difference of 20 minutes; Test type: Superiority or Other; p = 0.0077, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; This hierarchical, 2-sided testing procedure maintained the overall level of significance at approximately 0.05; Mean Difference (Net) = -9.153, 95% CI 2-sided [-15.857 to -2.448], Standard Error of Mean 2.422 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: WASO 1-8
Description: Wake Time After Sleep Onset, measured in minutes over the full 8 hour polysomnographic recording period, is summarized by treatment group for each night during the Screening and Treatment Periods.
Time Frame: Constantly throughout the 8 hour sleep period
Population: Intention to Treat population
Measure: Mean (Standard Error); unit: Minutes
Groups:
- Placebo: Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive placebo in place of the investigational zaleplon delayed and sustained release SKP-1041 tablets. Two placebo tablets were administered orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
Arm/Group | Placebo | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 67 | 67 | 67 | 67
Minutes | -44.65 (2.715) [-50.005 to -39.293] | -50.25 (2.755) [-55.688 to -44.819] | -51.56 (2.757) [56.999 to 46.123] | -50.17 (2.757)
Statistical Analysis 1: Comparison: Placebo vs 10 mg SKP-1041; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1476, Mixed Models Analysis — Adjusted mean differences were analyzed via general linear model that used change from baseline as response variable and included effects for patient, period, sequence, and treatment; No adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = -5.604, 95% CI 2-sided [-13.208 to 2.000], Standard Error of Mean 2.755 — A negative mean change from baseline indicates an improvement
Statistical Analysis 2: Comparison: Placebo vs 15 mg SKP-1041; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0757, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; No adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = -6.912, 95% CI 2-sided [-14.546 to 0.722], Standard Error of Mean 2.757 — A negative mean change from baseline indicates an improvement
Statistical Analysis 3: Comparison: Placebo vs 20 mg SKP-1041; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1553, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; No adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = -5.521, 95% CI 2-sided [-13.154 to 2.113], Standard Error of Mean 2.757 — A negative mean change from baseline indicates an improvement

3. Secondary Outcome: Total Sleep Time 3-7 Hours Post-dose
Description: Total Sleep Time during hours 3-7 (inclusive) post-dose
Time Frame: hours 3-7 (inclusive) post-dose
Population: Intention to Treat population (all randomized patients)
Measure: Mean (Standard Error); unit: Minutes
Groups:
- Placebo (Sugar Pill): Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive placebo in place of the investigational zaleplon delayed and sustained release SKP-1041 tablets. Two placebo tablets were administered orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
Arm/Group | Placebo (Sugar Pill) | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 67 | 67 | 67 | 67
Minutes | 39.03 (2.365) | 47.86 (2.400) | 49.46 (2.401) | 49.18 (2.402)
Statistical Analysis 1: Comparison: Placebo (Sugar Pill) vs 10 mg SKP-1041; The adjusted mean differences were analyzed by using a general linear model that used change from baseline as the response variable and included effects for patient, period, sequence, and treatment; Test type: Superiority or Other; p = 0.0092, Mixed Models Analysis — All aspects of the study's primary endpoint were statistically significant, and no adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = 8.831, 95% CI 2-sided [2.208 to 15.454], Standard Error of Mean 2.400 — A positive mean difference from baseline indicates an improvement
Statistical Analysis 2: Comparison: Placebo (Sugar Pill) vs 15 mg SKP-1041; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 10.425, 95% CI 2-sided [3.775 to 17.075], Standard Error of Mean 2.402 — A positive mean difference from baseline indicates an improvement
Statistical Analysis 3: Comparison: Placebo (Sugar Pill) vs 20 mg SKP-1041; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 10.147, 95% CI 2-sided [3.498 to 16.796], Standard Error of Mean 2.402 — A positive mean difference from baseline indicates an improvement

4. Secondary Outcome: Number of Awakenings After Sleep Onset During Hours 3 to 7 Post-dose (NAASO 3-7)
Description: Number of Awakenings After Sleep Onset during hours 3-7 post-dose (inclusive) as measured with PSG (polysomnography)
Time Frame: hours 3-7 (inclusive) post-dose
Population: Intention to Treat dataset (all randomized patients)
Measure: Mean (Standard Error); unit: Number of awakenings
Arm/Group | Placebo | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 67 | 67 | 67 | 67
Number of awakenings | -1.40 (0.240) | -1.96 (0.244) | -2.43 (0.244) | -2.19 (0.244)
Statistical Analysis 1: Comparison: Placebo vs 10 mg SKP-1041; This endpoint summarizes the number of times during Hours 3 7, after onset of persistent sleep, that there was a wake entry of at least 2 epochs duration. To be counted, each entry must have been separated by a sleep stage of 2, 3 4, or rapid eye movement; Test type: Superiority or Other; p = 0.1005, Mixed Models Analysis — Adjusted mean differences were analyzed with a general linear model that used change from baseline as the response variable and included effects for patient, period,sequence, and treatment; No adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = -0.562, 95% CI 2-sided [-1.235 to 0.110], Standard Error of Mean 0.244 — A negative mean change from baseline indicates an improvement
Statistical Analysis 2: Comparison: Placebo vs 15 mg SKP-1041; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; No adjustment for multiple testing was made for secondary endpoints; Mean Difference (Net) = -1.037, 95% CI 2-sided [-1.712 to -0.362], Standard Error of Mean 0.244 — A negative mean change from baseline indicates an improvement
Statistical Analysis 3: Comparison: Placebo vs 20 mg SKP-1041; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0216, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; No adjustments for multiple testing were made for secondary efficacy endpoints; Mean Difference (Net) = -0.793, 95% CI 2-sided [-1.467 to -0.118], Standard Error of Mean 0.244 — A negative mean change from baseline indicates an improvement

5. Secondary Outcome: Subjective Wake Time After Sleep Onset (sWASO)
Description: Subjective wake time after sleep onset sourced from the Morning Sleep Questionnaire self-assessment
Time Frame: 9 hours after tablet ingestion
Population: All Efficacy Analyses were performed on the Intention to Treat (ITT) population (all randomized patients).
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 67 | 67 | 67 | 67
minutes | -14.05 (4.873) | -22.50 (4.869) | -12.68 (4.937) | -25.89 (4.936)
Statistical Analysis 1: Comparison: Placebo vs 10 mg SKP-1041; Study was powered on the primary endpoint. Data for sWASO were sourced from Question 5 of the Morning Sleep Questionnaire. Its analysis follows a general linear model change from baseline as response variable including effects for patient, period, sequence, and treatment; Test type: Superiority or Other; p = 0.2190, Mixed Models Analysis — Mean (SEM) = adjusted mean change from baseline in each group (and standard error of the mean) and P value = P value for the comparison of the SEM of the active group with that of the placebo group; No adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = -8.452, 95% CI 2-sided [-21.980 to 5.077], Standard Error of Mean 0.2190 — A negative mean change from baseline indicates an improvement
Statistical Analysis 2: Comparison: Placebo vs 15 mg SKP-1041; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.8441, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; No adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = 1.365, 95% CI 2-sided [-12.327 to 15.056], Standard Error of Mean 4.937 — A positive mean change from baseline indicates a worsening
Statistical Analysis 3: Comparison: Placebo vs 20 mg SKP-1041; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0894, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; No adjustment for multiple testing was made for secondary efficacy endpoints; Mean Difference (Net) = -11.840, 95% CI 2-sided [-25.522 to 1.842], Standard Error of Mean 4.936 — A negative mean change from baseline indicates an improvement

6. Secondary Outcome: Digit Symbol Substitution Test
Description: Assessment of next-day residual cognitive effects. The Digit Symbol Substitution Test (DSST) explores attention and psychomotor speed. Given a code table displaying the correspondence between pairs of digits (from 1 to 9) and symbols, the patient filled in blank squares with the symbol that was paired with the digit displayed above the square. The patient was required to fill in as many squares as possible in 180 seconds.
Time Frame: 9 hours after tablet ingestion
Population: Intention to Treat population (all randomized patients)
Measure: Mean (Standard Error); unit: percentage change from mean baseline
Arm/Group | Placebo | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 67 | 67 | 67 | 67
percentage change from mean baseline | 8.56 (1.434) | 9.26 (1.469) | 6.59 (1.523) | 9.95 (1.626)
Statistical Analysis 1: Comparison: Placebo vs 10 mg SKP-1041; Adjusted mean differences were analyzed by using a general linear model that used change from baseline as the response variable; Test type: Superiority or Other; p = 0.6433, Mixed Models Analysis — Analysis included effects for patient, period, sequence and treatment; Mean Difference (Net) = 0.560, 95% CI 2-sided [-1.823 to 2.943], Standard Error of Mean 1.469 — A positive mean difference from baseline indicates improvement
Statistical Analysis 2: Comparison: Placebo vs 15 mg SKP-1041; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1167, Mixed Models Analysis — Analysis included effects for patient, period, sequence and treatment; Mean Difference (Net) = -1.912, 95% CI 2-sided [-4.304 to 0.481], Standard Error of Mean 1.523 — A negative mean difference from baseline indicates a worsening
Statistical Analysis 3: Comparison: Placebo vs 20 mg SKP-1041; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.2385, Mixed Models Analysis — Analysis included effects for patient, period, sequence and treatment; Mean Difference (Net) = 1.434, 95% CI 2-sided [-0.958 to 3.826], Standard Error of Mean 1.626 — A positive mean difference from baseline indicates improvement

7. Secondary Outcome: Digit Span Test
Description: Assessment of next day residual cognitive effects via testing immediate recall of numbers. The patient was given a string of digits and asked to repeat them forward, and then a second string of digits to repeat backward. The score was the number of correct responses, where the digits were repeated correctly. One point was given for each correctly repeated string of digits. The maximum subscore in the Digits Forward was 16, and the maximum subscore in the Digits Backward was 14, for a total score of 30.
Time Frame: 9 hours post-dose
Population: Intention to Treat population (all randomized patients)
Measure: Mean (Standard Error); unit: units on a scale change from baseline
Groups:
- 10 mg SKP=1041: Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive 10mg of the investigational zaleplon delayed and sustained release SKP-1041 tablets. One 10 mg SKP-1041 tablet and one placebo tablet were administered orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
Arm/Group | Placebo | 10 mg SKP=1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 67 | 67 | 67 | 67
units on a scale change from baseline | 0.23 (0.268) | 0.71 (0.256) | 0.40 (0.259) | -0.02 (0.237)
Statistical Analysis 1: Comparison: Placebo vs 10 mg SKP=1041; The adjusted mean differences were analyzed with a general linear model that used change from baseline as the response variable and included effects for patient, period, sequence and treatment; Test type: Superiority or Other; p = 0.0914, Mixed Models Analysis; Mean Difference (Net) = 0.450, 95% CI 2-sided [-0.073 to 0.972], Standard Error of Mean 0.256 — A positive mean change from baseline indicates an improvement
Statistical Analysis 2: Comparison: Placebo vs 15 mg SKP-1041; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.5360, Mixed Models Analysis; Mean Difference (Net) = 0.165, 95% CI 2-sided [-0.360 to 0.690], Standard Error of Mean 0.259 — A positive mean change from baseline indicates an improvement
Statistical Analysis 3: Comparison: Placebo vs 20 mg SKP-1041; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.3254, Mixed Models Analysis; Mean Difference (Net) = -0.262, 95% CI 2-sided [-0.787 to 0.263], Standard Error of Mean 0.237 — A negative mean change from baseline indicates a worsening

8. Secondary Outcome: Visual Analog Scale (Sedation)
Description: Self-assessment of next morning sedation. Patients answered the question "How alert do you feel?" via a 100mm scale on which 0mm indicated "very sleepy" and 100mm indicated "wide awake and alert".The VAS measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Operationally, a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end (in this case, sleepiness and alertness). Patients were asked to mark the point on the line that they felt represented their current state. The VAS score was determined by measuring in millimeters from the left-hand end of the line to the point that the patient marked.
Time Frame: 9 hours after tablet ingestion
Population: Safety population (patients exposed to that given treatment)
Measure: Mean (Standard Error); unit: mm change from baseline
Groups:
- 10 mg SKP-1041: Each patient was assigned at some point in their randomized crossover sequence of four treatment arms to receive 10 mg of the investigational zaleplon delayed and sustained release SKP-1041 tablets. One 10 mg SKP-1041 tablet and one placebo tablet were administered orally at bedtime for each of two consecutive nights during the Sleep Study. Afterward, patients were released from the sleep laboratory, washed out at home for 4-7 days, and returned to the sleep lab for the next treatment in their randomized sequence.
Arm/Group | Placebo (Sugar Pill) | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 66 | 65 | 65 | 65
mm change from baseline | 3.48 (2.195) | 3.83 (1.818) | 3.55 (2.422) | 4.96 (2.058)
Statistical Analysis 1: Comparison: Placebo (Sugar Pill) vs 10 mg SKP-1041; Test type: Superiority or Other; p = 0.7190, Mixed Models Analysis — Adjusted mean differences were analyzed in a general linear model that used change from baseline as the response variable; The Model included effects for patient, period, sequence and treatment; Mean Difference (Net) = 0.710, 95% CI 2-sided [-3.175 to 4.595], Standard Error of Mean 1.818 — A positive mean change from baseline indicates improvement
Statistical Analysis 2: Comparison: Placebo (Sugar Pill) vs 15 mg SKP-1041; Test type: Superiority or Other; p = 0.6784, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; The Model included effects for patient, period, sequence and treatment; Mean Difference (Net) = 0.821, 95% CI 2-sided [-3.080 to 4.722], Standard Error of Mean 2.422 — A positive mean change from baseline indicates an improvement
Statistical Analysis 3: Comparison: Placebo (Sugar Pill) vs 20 mg SKP-1041; Test type: Superiority or Other; p = 0.2433, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; The Model included effects for patient, period, sequence and treatment; Mean Difference (Net) = 2.314, 95% CI 2-sided [-1.586 to 6.214], Standard Error of Mean 2.058 — A positive mean change from baseline indicates an improvement

9. Secondary Outcome: Cmax Pharmacokinetic (PK) Profile Characterization
Description: A detailed characterization of the Cmax (maximum plasma concentration of SKP-1041 zaleplon in ng/mL) for each of the 3 study doses within the Pharmacokinetic Population (patients who completed the PK substudy--night 3 of Visit 6)with subsequent descriptive statistics comparing key PK characteristics across the 3 doses.
  Descriptive statistics and analysis of variance (ANOVA) for independent groups compared the three dosage groups using the untransformed values, as well as following rank transformation(nonparametric analysis).
Time Frame: Blood samples drawn hourly from -1 to 10 hours post-dose (except hour 7)
Population: Pharmacokinetic Population--Patients who completed night 3 of Visit 6 (the PK substudy). Note that these patients had participated in a crossover design across all doses for the sleep study but had PK assessments only for one dose (parallel group design).
Measure: Mean (Standard Error); unit: ng/mL
Units Other Than Participants: Blood samples
Groups:
- 10 mg SKP-1041: The fourth and final treatment period included a third night at the site during which all patients continued to receive the same study medication as on the first 2 nights of this treatment period. Patients randomized to this group were administered one placebo and one 10 mg SKP-1041 tablet at bedtime for the third time. Blood was drawn from all patients for PK analyses at specific time intervals.
- 15 mg SKP-1041: The fourth and final treatment period included a third night at the site during which all patients continued to receive the same study medication as on the first 2 nights of this treatment period. Patients randomized to this group were administered one placebo and one 15 mg SKP-1041 tablet at bedtime for the third time. Blood was drawn from all patients for PK analyses at specific time intervals.
- 20 mg SKP-1041: The fourth and final treatment period included a third night at the site during which all patients continued to receive the same study medication as on the first 2 nights of this treatment period. Patients randomized to this group were administered two 10 mg SKP-1041 tablets at bedtime for the third time. Blood was drawn from all patients for PK analyses at specific time intervals.
Arm/Group | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 17 | 13 | 15
Number analyzed (Blood samples) | 170 | 130 | 150
ng/mL | 17.9 (1.3) | 25.3 (2.9) | 34.4 (4.2)
Statistical Analysis 1: Comparison: 10 mg SKP-1041 vs 15 mg SKP-1041 vs 20 mg SKP-1041; Cmax(ng/mL) [Maximum plasma zaleplon concentration]; Test type: Superiority or Other; p = 0.0009, ANOVA; F-test 2 degrees of freedom; Mean Difference (Net) = 8.39

10. Secondary Outcome: Cmax/Dose(Dose-Normalized Cmax)Pharmacokinetic (PK) Profile Characterization
Description: A detailed characterization of Cmax/Dose (ng/mL/mg) (maximum plasma zaleplon concentration normalized per dose) PK profile of SKP-1041 zaleplon for each of the 3 study doses within the Pharmacokinetic Population (patients who completed the PK substudy--night 3 of Visit 6)with subsequent descriptive statistics comparing key PK characteristics across the 3 doses.
  Descriptive statistics, geometric means and 90% confidence intervals were calculated for dose-normalized values of Cmax. Analysis of variance (ANOVA) for independent groups compared the three dosage groups using the untransformed values, as well as following rank transformation(nonparametric analysis).
Time Frame: Blood samples drawn hourly from -1 to 10 hours post-dose (except hour 7)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: ng/mL/mg zaleplon
Units Other Than Participants: Blood Samples
Arm/Group | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 17 | 13 | 15
Number analyzed (Blood Samples) | 170 | 130 | 150
ng/mL/mg zaleplon | 1.8 (0.1) | 1.7 (0.2) | 1.7 (0.2)
Statistical Analysis 1: Comparison: 10 mg SKP-1041 vs 15 mg SKP-1041 vs 20 mg SKP-1041; Cmax normalized per dose; Test type: Superiority or Other; p = 0.9142, ANOVA; F-test two degrees of freedom; Mean Difference (Net) = 0.09

11. Secondary Outcome: Tmax Pharmacokinetic (PK) Profile Characterization
Description: A detailed characterization of Tmax (hour) (timepoint post-dose of maximum plasma zaleplon concentration) PK profile of SKP-1041 zaleplon for each of the 3 study doses within the Pharmacokinetic Population (patients who completed the PK substudy--night 3 of Visit 6)with subsequent descriptive statistics comparing key PK characteristics across the 3 doses.
  Descriptive statistics and analysis of variance (ANOVA) for independent groups compared the three dosage groups using the untransformed values, as well as following rank transformation(nonparametric analysis).
Time Frame: Blood samples drawn hourly from -1 to 10 hours post-dose (except hour 7)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: Hours post-dose
Units Other Than Participants: Blood Samples
Arm/Group | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 17 | 13 | 15
Number analyzed (Blood Samples) | 170 | 130 | 150
Hours post-dose | 4 (2.5) | 4 (2.5) | 4 (3.6)
Statistical Analysis 1: Comparison: 10 mg SKP-1041 vs 15 mg SKP-1041 vs 20 mg SKP-1041; Time (hour)post-dose of maximum plasma zaleplon concentration; Test type: Superiority or Other; p = 0.1193, ANOVA; F-test 2 degrees of freedom; Mean Difference (Net) = 2.24

12. Secondary Outcome: AUC Pharmacokinetic (PK) Profile Characterization
Description: A detailed characterization of the AUC (area under the concentration-time curve of SKP-1041 zaleplon) for each of the 3 study doses within the Pharmacokinetic Population (patients who completed the PK substudy--night 3 of Visit 6)with subsequent descriptive statistics comparing key PK characteristics across the 3 doses.
  Descriptive statistics were calculated for AUC. Analysis of variance (ANOVA) for independent groups compared the three dosage groups using the untransformed values, as well as following rank transformation(nonparametric analysis).
Time Frame: Blood samples drawn hourly from -1 to 10 hours post-dose (except hour 7)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: ng x h/mL
Units Other Than Participants: Blood Samples
Arm/Group | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 17 | 13 | 15
Number analyzed (Blood Samples) | 170 | 130 | 150
ng x h/mL | 56.5 (3.9) | 77.4 (5.6) | 135.3 (22.0)
Statistical Analysis 1: Comparison: 10 mg SKP-1041 vs 15 mg SKP-1041 vs 20 mg SKP-1041; AUC ng*h/mL); Test type: Superiority or Other; p = 0.0003, ANOVA; F-test 2 degrees of freedom; Mean Difference (Net) = 9.85

13. Secondary Outcome: AUC/Dose (ng*h/mL/mg) Pharmacokinetic (PK) Profile Characterization
Description: A detailed characterization of the AUC/Dose (ng*h/mL/mg) [Area under the concentration-time curve per Dose of SKP-1041 zaleplon] for each of the 3 study doses within the Pharmacokinetic Population (patients who completed the PK substudy--night 3 of Visit 6)with subsequent descriptive statistics comparing key PK characteristics across the 3 doses.
  Descriptive statistics and analysis of variance (ANOVA) for independent groups compared the three dosage groups using the untransformed values, as well as following rank transformation(nonparametric analysis).
Time Frame: Blood samples drawn hourly from -1 to 10 hours post-dose (except hour 7)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: ng*h/mL/mg
Units Other Than Participants: Blood Samples
Arm/Group | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 17 | 13 | 15
Number analyzed (Blood Samples) | 170 | 130 | 150
ng*h/mL/mg | 5.36 (0.4) | 5.20 (0.4) | 6.76 (1.1)
Statistical Analysis 1: Comparison: 10 mg SKP-1041 vs 15 mg SKP-1041 vs 20 mg SKP-1041; AUC/Dose (ng*h/mL/mg); Test type: Superiority or Other; p = 0.2281, ANOVA; F-test 2 degrees of freedom; Mean Difference (Net) = 1.28

14. Secondary Outcome: Half-Life (t1/2 Hour) Pharmacokinetic (PK) Profile Characterization
Description: A detailed characterization of the plasma Half-Life (t1/2 in hours) of SKP-1041 zaleplon the each of the 3 study doses within the Pharmacokinetic Population (patients who completed the PK substudy--night 3 of Visit 6)with subsequent descriptive statistics comparing key PK characteristics across the 3 doses.
  Descriptive statistics and analysis of variance (ANOVA)for independent groups compared the three dosage groups using the untransformed values, as well as following rank transformation(nonparametric analysis).
Time Frame: Blood samples drawn hourly from -1 to 10 hours post-dose (except hour 7)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: hour
Units Other Than Participants: Blood Samples
Arm/Group | 10 mg SKP-1041 | 15 mg SKP-1041 | 20 mg SKP-1041
Number analyzed (Participants) | 17 | 13 | 15
Number analyzed (Blood Samples) | 170 | 130 | 150
hour | 1.52 (0.05) | 1.65 (0.17) | 1.47 (0.09)
Statistical Analysis 1: Comparison: 10 mg SKP-1041 vs 15 mg SKP-1041 vs 20 mg SKP-1041; Half-Life (t1/2 in hours) of plasma zaleplon from each of 3 doses of SKP-1041; Test type: Superiority or Other; p = 0.4835, ANOVA; 2 degrees of freedom F-test; Mean Difference (Net) = 0.74

ADVERSE EVENTS:
Time Frame: 6 months
Description: 21 patients (31.3%) reported at least 1 Treatment Emergent Adverse Event (TEAE), 6 of whom (9.0%) experienced at least 1 TEAE that was considered related to study medication. All TEAEs were mild or moderate in intensity. There were no Serious AEs,no TEAEs leading to discontinuation of study medication, and no TEAEs that led to death.
Groups:
- Placebo; 10 mg; 15mg; 20mg: Each of the 67 patients was randomly assigned a sequence of the four treatment arms, washed out, and then crossed over to the next assigned treatment in their sequence.
Arm/Group | Placebo | 10 mg | 15mg | 20mg
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 6/67 | 7/67 | 9/67 | 7/67
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=67) | 10 mg (N=67) | 15mg (N=67) | 20mg (N=67)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion Site Haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Questionnaires focused on initial insomnia as opposed to middle of the night awakening, short exposure to each dose, and lengthy washout periods between doses, may not allow for ideal assessment of subjective response to treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PROTOCOL CONFIDENTIALITY/COMPLIANCE STATEMENT:

Investigators "...agree not to originate or use the name of Somnus Therapeutics, Inc and/or Zaleplon or SKP-1041, or any of its employees, in any publicity, news release, or other public announcement, written or oral, whether to the public, press, or otherwise, relating to this protocol, to any amendment hereto, or to the performance hereunder, without the prior written consent of Somnus Therapeutics, Inc."

"SKP" refers to SkyePharma PLC